CLINICAL TRIAL: NCT05530226
Title: A Single Arm Study of Traditional Chinese Medicine for Treatment of Plasma Cell Mastitis
Brief Title: A Single Arm Study of Traditional Chinese Medicine for Plasma Cell Mastitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Professor, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LCG013
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Plasma Cell Mastitis
MeSH Terms: interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Intervention Model Description: single arm study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traditional Chinese medicine group (Experimental): Traditional Chinese medicine, twice daily
  Interventions: Drug: Traditional Chinese medicine

INTERVENTIONS:
Drug: Traditional Chinese medicine — Traditional Chinese medicine, oral administration, twice daily
  Other Names: Traditional herbal medicine

SUMMARY:
This is a single-center, single-arm, open-label trial evaluating the efficacy and safety of traditional Chinese medicine for plasma cell mastitis.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label trial evaluating the efficacy and safety of traditional Chinese medicine for plasma cell mastitis. This study will include 50 patients with plasma cell mastitis. After providing written informed consent, the participants will receive traditional herbal medicine twice daily. Efficacy will be assessed every 15 days. If the disease progresses, the participant will withdraw from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for plasma cell mastitis.
2. Women aged > 20 years and ≤ 60 years.
3. Karnofsky Performance Status (KPS) Scale score ≥ 70.
4. Volunteers to participate in the study, provision of signed informed consent, good compliance and willingness to cooperate with follow-ups.

Exclusion Criteria:

1. Pregnant and lactating women; fertile women who provide positive results of baseline pregnancy test; women of childbearing age who are unwilling to take effective contraceptive measures during the whole study period.
2. Patients with serious underlying diseases, such as diabetes, cardiovascular and cerebrovascular diseases, liver, kidney and hematopoietic system diseases.
3. Allergic constitution, such as a history of allergies to two or more drugs or foods; or those who are known to be allergic to the ingredients of the drugs used in this trial.
4. Recent use of antidepressants and other psychotropic drugs.
5. Hormone and immunosuppressive therapy were used one month before enrollment.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | During treatment（1 month to 6 months）
  the proportion of patients who completely respond to the treatment at any study time point
Clinical response rate | During treatment（1 month to 6 months）
  the proportion of patients who respond to the treatment at any study time point

SECONDARY OUTCOMES:
Surgical rate | During treatment（1 month to 6 months）
  the proportion of patients who receive surgery at any study time point
Local recurrence rate | Within 6 months after treatment
  the proportion of patients who recur at any study time point
Adverse events (AE) and serious adverse events (SAE) | During treatment（1 month to 6 months）
  For adverse events (AE) and serious adverse events (SAE), refer to NCI-CTC AE 5.0 standard.

OTHER OUTCOMES:
Expression of immune cells | During treatment（1 month to 6 months）
  Expression of immune cells (T cell, B cell, NK cell)
Expression of cytokines (IL, INF-r, TNF-a) | During treatment（1 month to 6 months）
  Expression of cytokines (IL, INF-r, TNF-a)
C-reactive protein | During treatment（1 month to 6 months）
  Expression of c-reactive protein
Clinical symptom scores | During treatment（1 month to 6 months）
  Clinical symptom scores were measured using traditional Chinese medicine clinical symptom assessment with reference to The Disease Diagnosis Curative Effect of Traditional Chinese Medicine Standard. The clinical symptom scales include mass size, swelling, discharge, retraction, abscess, fistula. The higher the score, the worse the symptom. Clinical symptom scores of patients before and after treatment were observed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Liu C, Yu H, Chen G, Yang Q, Wang Z, Niu N, Han L, Zhao D, Wang M, Liu Y, Yang Y. An herbal drug combination identified by knowledge graph alleviates the clinical symptoms of plasma cell mastitis patients: A nonrandomized controlled trial. Elife. 2023 Mar 14;12:e84414. doi: 10.7554/eLife.84414. PMID 36917037